CLINICAL TRIAL: NCT06373861
Title: Generating Advancements Through Longitudinal Analysis in X and Y Variations
Brief Title: Generating Advancements Through Longitudinal Analysis in X and Y Variations (GALAXY)
Acronym: GALAXY
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0482
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Sex Chromosome Aneuploidy
Keywords: X&Y variations; chromosome variations; Klinefelter; XXY; XXX; XYY; tetrasomy; pentasomy; trisomy
MeSH Terms: conditions — Klinefelter Syndrome; Tetrasomy; Trisomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — If resources are available and optional consent is provided, a 5-10mL blood sample will be obtained in 1 gold top and 1 purple top (EDTA) tube and processed for storage of plasma, serum, and buffy coat. These specimens will be stored in a biobank with a barcode to link the sample with the patient for future studies involving the assessment of hormones, proteins, metabolites, DNA, RNA, and other studies. Phlebotomy will be combined with clinical phlebotomy whenever possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — This study is an observational study without treatment intervention.

SUMMARY:
GALAXY is a registry research study that plans to learn more about individuals with X&Y variations (also called sex chromosome aneuploidies) through collecting information from medical records.This includes genetic tests, imaging, medications, and more for hundreds of patients seen at a number of clinics across the US. The purpose of the GALAXY Registry is to collect and store this information with the overall goal to improve health outcomes in individuals with X&Y variations and the care they receive.

ELIGIBILITY:
Inclusion Criteria:

1. Genetically-confirmed diagnosis of a sex chromosome aneuploidy condition
2. Any age
3. Any gender
4. Informed consent for individuals >18 years of age, parent/guardian permission for individuals <18 or proxy-consent from legally authorized representative if impaired decision making

Exclusion Criteria:

a. Lack of documentation of genetic testing confirming SCA diagnosis

Ages: 0 Days to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population for this registry is patients diagnosed with sex chromosome aneuploidy (SCA) conditions throughout the lifespan.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2037-04 (Estimated); Study Completion 2037-04 (Estimated)

PRIMARY OUTCOMES:
Health Conditions | From study start until condition observed, up to 15 years
  Average number of chronic diagnoses per person

SECONDARY OUTCOMES:
Prevalence of mental health diagnoses | From study start until condition observed, up to 15 years
  Prevalence of mental health diagnoses is defined as the number of participants in the sample diagnosed with a mental health disorder by a clinician according to their medical record out of the total sample. This will be determined by a diagnosis of any of the following in a clinical encounter, problem list, and/or past medical history:
  * Depression
  * Anxiety
  * Mood disorder NOS
  * Psychotic disorder
  * Attention-deficit/hyperactivity disorder (ADHD)
  * Autistic disorder
Cardiometabolic diagnoses - prevalence of obesity | From study start until condition observed, up to 15 years
  Prevalence of obesity is defined as the number of participants in the sample with obesity in their medical record out of the total sample. Obesity in pediatric populations is determined using BMI-for-age and obesity in adult populations is determined using BMI. BMI is calculated as the weight in kilograms divided by the height in meters squared.
  Participants will be considered to have obesity if:
  * There is a diagnosis of obesity in the medical record in a clinical encounter, problem list, and/or past medical history
  * For children 17 years and younger: there is an available growth chart/height/weight/other data necessary to calculate the BMI-for-age and the BMI-for-age is at or above the 95th percentile
  * For adults 18 years and older: there is a BMI at or above 30 kg/m2 or the data necessary to calculate BMI and it is at or above 30 kg/m2
Cardiometabolic diagnoses - prevalence of dyslipidemia | From study start until condition observed, up to 15 years
  Prevalence of metabolic syndrome is defined as the number of participants in the sample with dyslipidemia in their medical record out of the total sample. Dyslipidemia will be defined as:
  * Diagnosis of dyslipidemia, hypertriglyceridemia, hypercholesterolemia in a clinical encounter, problem list, and/or past medical history
  * Laboratory evidence of elevated total cholesterol, LDL, triglycerides, and/or low HDL for sex and age
Cardiometabolic diagnoses-prevalence of hypertension | From study start until condition observed, up to 15 years
  Prevalence of hypertension is defined as the number of participants in the sample with evidence of hypertension in their medical record out of the total sample. Evidence of hypertension includes:
  * Formal diagnosis of hypertension in a clinical encounter, problem list, and/or past medical history
  * For children under 13 years old: a blood pressure reading at or above the 95th percentile for age, height, and sex
  * For children between 13 and 17 years old: a blood pressure reading at or above 130/80 mmHg
  * For adults 18 years or older: a blood pressure reading at or above 140/90 mmHg
Autoimmune diagnoses - prevalence of hypothyroidism and of hyperthyroidism | From study start until condition observed, up to 15 years
  Prevalence of hypothyroidism is defined as the number of participants in the sample with evidence of hypertension in their medical record out of the total sample.
Autoimmune diagnoses - prevalence of diabetes | From study start until condition observed, up to 15 years
  Prevalence of diabetes is defined as the number of participants in the sample with evidence of hypertension in their medical record out of the total sample. Both type 1 and type 2 are included.

CONTACTS AND LOCATIONS:
Overall Officials: Shanlee M Davis, MD, PhD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States